CLINICAL TRIAL: NCT03603353
Title: Substudy of Efficacy, Safety and Toxicology of Electronic Nicotine Delivery Systems as an Aid for Smoking Cessation (ESTxENDS Trial)- the Sleep Quality Substudy of ESTxENDS
Brief Title: The ESTxENDS Trial- Substudy on the Effects of Using Electronic Nicotine Delivery Systems (ENDS) on Sleep Quality.
Acronym: ESTxENDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: University of Lausanne (Other); University of Geneva, Switzerland (Other); University of Zurich (Other); State Hospital, St. Gallen (Other Government); Swiss National Science Foundation (Other); Krebsforschung Schweiz, Bern, Switzerland (Other); Federal Office of Public Health, Switzerland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-02332g
Record Dates: First submitted 2018-07-02; First posted 2018-07-27 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Smoking Cessation; Sleep
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Masking Description: Statisticians and laboratory personnel will be blinded to group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: ENDS (vaporizer/e-cig) and smoking cessation counseling
- Control group (Active Comparator)
  Interventions: Other: Smoking cessation counseling

INTERVENTIONS:
Other: ENDS (vaporizer/e-cig) and smoking cessation counseling — Participants in the intervention group will receive an ENDS and nicotine-containing e-liquids, which they will be allowed to use ad libitum. Additionally, they will receive smoking cessation counseling.
  Participants will be allowed to additionally use nicotine replacement therapy. All participants will be followed over a 24-month period. Smoking cessation counseling will be provided in person at the first clinical visit and then over the phone at the target quit date one week later and again at week 2, 4 and 8 after the target quit date. After 6, 12 and 24 months, participants will be asked to come to a clinical visit.
  Arms: Intervention group
Other: Smoking cessation counseling — Participants in the control group will receive smoking cessation counseling only. Participants will be allowed to additionally use nicotine replacement therapy. All participants will be followed over a 24-month period. Smoking cessation counseling will be provided in person at the first clinical visit and then over the phone at the target quit date one week later and again at week 2, 4 and 8 after the target quit date. After 6, 12 and 24 months, participants will be asked to come to a clinical visit.
  Arms: Control group

SUMMARY:
--> This is a substudy of the main ESTxENDS trial (NCT03589989). Sleep quality outcomes should be considered secondary outcomes of the main smoking cessation outcome formulated in NCT03589989.

Cigarette smoking is the leading cause of preventable death in Switzerland and still more than a quarter of the Swiss population smokes cigarettes. Recently, electronic nicotine delivery systems (ENDS; also called vaporizer or electronic cigarette) have become popular with smokers who want to stop smoking or reduce their exposure to inhaled chemicals since ENDS use appears to be safer than tobacco smoking.

The majority of attempts to quit tobacco smoking do not end in success due to unpleasant withdrawal symptoms. One of such symptoms is disturbed sleep. Sleep disturbances are a problem for smokers who are trying to quit. Sleep disturbances results from difficulty falling asleep or frequent arousals after sleep onset, and have negative daytime consequences such as sleepiness and dysphoric mood. Studies indicate that awakenings during night affect the cardiovascular system by providing repetitive bursts of sympathetic nervous system activation, likely contributing to elevated levels of cardiovascular and cerebrovascular morbidity. ENDS with nicotine containing e-liquids may be effective in assisting with tobacco smoking cessation by reducing withdrawal-induced sleep disturbances.

This study will therefore test the efficacy of ENDS for cigarette smoking cessation, the safety of ENDS on adverse events and the effect of ENDS on health-related outcomes and exposure to inhaled chemicals.

For the main ESTxENDS trial (NCT03589989), cigarette smokers motivated to quit smoking cigarettes will be included. Participants in the intervention group will receive an ENDS and nicotine-containing e-liquids, which they will be allowed to use ad libitum. Additionally, they will receive smoking cessation counseling. Participants in the control group will receive smoking cessation counseling only. All participants will be followed over a 24-month period. Sleep quality will be assessed using the Pittsburgh sleep quality index- questionnaire at baseline and at 6, 12 and 24 months' follow-up.

ELIGIBILITY:
Inclusion criteria:

* Informed Consent as documented by signature
* Persons aged 18 or older
* Currently smoking 5 or more cigarettes a day for at least 12 months
* Willing to try to quit smoking within the next 3 months,
* Persons providing a valid phone number, a valid email address and/or a valid postal address.

Exclusion criteria:

* Known hypersensitivity or allergy to contents of the e-liquid
* Participation in another study with investigational drug within the 30 days preceding the baseline visit and during the present study where interactions are to be expected
* Women who are pregnant or breast feeding
* Intention to become pregnant during the course of the scheduled study intervention, i.e. within the first 6-months of the study
* Persons having used ENDS or tobacco heating systems regularly in the 3 months preceding the baseline visit
* Persons having used nicotine replacement therapy (NRT) or other medications with demonstrated efficacy as an aid for smoking cessation such as varenicline or bupropion within the 3 months preceding the baseline visit
* Persons who cannot attend the 6- month follow-up visit for any reason
* Cannot understand instructions delivered in person or by phone, or otherwise unable to participate in study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1246 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Subjective sleep quality_1 | 6 months post quit date
  Subjective sleep quality assessed with the Pittsburgh Sleep Quality Index (PSQI).
Subjective sleep quality_2 | 12 months post quit date
  Subjective sleep quality assessed with the Pittsburgh Sleep Quality Index (PSQI).
Subjective sleep quality_3 | 24 months post quit date
  Subjective sleep quality assessed with the Pittsburgh Sleep Quality Index (PSQI).

SECONDARY OUTCOMES:
Change in subjective sleep quality | Change from baseline to 6,12, 24 months post quit date
  Subjective sleep quality assessed with the Pittsburgh Sleep Quality Index (PSQI).

CONTACTS AND LOCATIONS:
Overall Officials: Reto Auer, Prof.Dr.med, Study Director — Berner Institut für Hausarztmedizin (BIHAM); Micheline Maire, Dr., Study Director — Berner Institut für Hausarztmedizin (BIHAM)
Locations (5):
- Switzerland (5):
  - Unisanté, Centre universitaire de médecine générale et santé publique, Université de Lausanne, Lausanne, Canton of Vaud
  - University Clinic for General Internal Medicine, Bern University Hospital, Bern
  - Département de médecine interne, Hôpitaux universitaires de Genève, Geneva
  - Lungenzentrum, Klinik für Pneumologie und Schlafmedizin, Kantonsspital St. Gallen, Sankt Gallen
  - Epidemiology, Biostatistics and Prevention Institute (EBPI), University of Zurich, Zurich

REFERENCES:
- [Background] Hughes JR. Effects of abstinence from tobacco: etiology, animal models, epidemiology, and significance: a subjective review. Nicotine Tob Res. 2007 Mar;9(3):329-39. doi: 10.1080/14622200701188927. PMID 17365765
- [Background] Hughes JR, Higgins ST, Bickel WK. Nicotine withdrawal versus other drug withdrawal syndromes: similarities and dissimilarities. Addiction. 1994 Nov;89(11):1461-70. doi: 10.1111/j.1360-0443.1994.tb03744.x. PMID 7841857
- [Background] Wetter DW, Young TB. The relation between cigarette smoking and sleep disturbance. Prev Med. 1994 May;23(3):328-34. doi: 10.1006/pmed.1994.1046. PMID 8078854
- [Background] Colrain IM, Trinder J, Swan GE. The impact of smoking cessation on objective and subjective markers of sleep: review, synthesis, and recommendations. Nicotine Tob Res. 2004 Dec;6(6):913-25. doi: 10.1080/14622200412331324938. PMID 15801567
- [Background] Bertrand D. The possible contribution of neuronal nicotinic acetylcholine receptors in depression. Dialogues Clin Neurosci. 2005;7(3):207-16. doi: 10.31887/DCNS.2005.7.3/dbertrand. PMID 16156379
- [Background] Grandner MA, Jackson NJ, Pak VM, Gehrman PR. Sleep disturbance is associated with cardiovascular and metabolic disorders. J Sleep Res. 2012 Aug;21(4):427-33. doi: 10.1111/j.1365-2869.2011.00990.x. Epub 2011 Dec 12. PMID 22151079